CLINICAL TRIAL: NCT00964379
Title: Prospective Randomized Trial of Intraperitoneal Versus Extraperitoneal Techniques for Construction of Terminal Iliac Fossa Colostomies
Brief Title: Intraperitoneal Versus Extraperitoneal Colostomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Bruce G. Wolff, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 528-93
Record Dates: First submitted 2009-08-11; First posted 2009-08-24 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Colostomy
Keywords: Intra versus extraperitoneal colostomy
MeSH Terms: interventions — Infusions, Parenteral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intraperitoneal colostomy (Active Comparator)
  Interventions: Procedure: intraperitoneal or extraperitoneal colostomy
- extraperitoneal colostomy (Active Comparator)
  Interventions: Procedure: intraperitoneal or extraperitoneal colostomy

INTERVENTIONS:
Procedure: intraperitoneal or extraperitoneal colostomy — creation of colostomy

SUMMARY:
This is a prospective randomized trial of intraperitoneal versus extraperitoneal techniques for construction of terminal iliac fossa colostomies.

ELIGIBILITY:
Inclusion Criteria:

* permanent colostomy

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 1988-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
parastomal hernia, stoma dysfunction | 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States